CLINICAL TRIAL: NCT02432807
Title: A Randomized, Multicenter, Double-Masked, Placebo-Controlled, Phase 3 Study to Evaluate the Safety and Efficacy of Vancomycin Hydrochloride Ophthalmic Ointment 1.1% in Patients With Moderate to Severe Bacterial Conjunctivitis
Brief Title: Safety and Efficacy of Vancomycin Ophthalmic Ointment in Patients With Moderate to Severe Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kurobe LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUR-1301-101
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin 1.1% (Experimental): Vancomycin hydrochloride ophthalmic ointment 1.1% dosed approximately 1 cm of ointment QID for 7 days
  Interventions: Drug: Vancomycin 1.1%
- Placebo (Placebo Comparator): Vehicle (placebo) ophthalmic ointment dosed approximately 1 cm of ointment QID for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin 1.1% — Vancomycin hydrochloride ophthalmic ointment 1.1%
  Arms: Vancomycin 1.1%
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3 study to evaluate the safety and efficacy of a vancomycin hydrochloride ophthalmic ointment dosed 4 times daily for 7 days compared to placebo (vehicle) in patients with moderate to severed Gram-positive bacterial conjunctivitis.

DETAILED DESCRIPTION:
Bacterial conjunctivitis is common ocular disease caused by various types of bacteria including methicillin-resistant Staphylococcus aureus (MRSA) and methicillin-resistant Staphylococcus epidermidis (MRSE). External ocular infections such as those caused by MRSA or MRSE frequently are not serious but in rare cases may be severe enough to threaten vision. When ocular infections due to resistant organisms such as MRSA/MRSE do not respond to empiric treatment with approved antibiotics, there are few treatment options. Vancomycin is one of the few treatment options that has been shown to be effective against all clinical isolates of MRSA/MRSE.

This study is a Phase 3 study to evaluate the safety and efficacy of a vancomycin hydrochloride ophthalmic ointment in patients with moderate to severed Gram-positive bacterial conjunctivitis including those with MRSA and MRSE. Subjects, who are adenovirus negative, will be dosed with vancomycin hydrochloride ophthalmic ointment or placebo (vehicle) 4 times daily for 7 days and evaluated for clinical and bacterial resolution of their infection along with an assessment of the safety of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 and older
2. Clinical diagnosis of acute bacterial conjunctivitis with at least one eye exhibiting conjunctival discharge graded ≥ 2 as well as palpebral conjunctival injection graded ≥ 2 AND bulbar conjunctival injection graded ≥ 2 with onset ≤ 4 days as reported by the subject.
3. Negative test result on AdenoPlus® adenovirus test.
4. Snellen visual acuity (VA) equal to or better than 20/200 in each eye using current corrective lenses, if required (or if worn) and/or using pinhole if subject's corrective lenses are not available at the time of exam. Every attempt should be made to obtain a VA measurement in children and, if it is unobtainable, the decision as to whether the criterion is met will be at the investigator's discretion.
5. Female subjects must be 1-year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Visit 1. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
6. Able to self-administer study medication or to have the study medication administered by a caregiver throughout the study period.
7. Must have signed written consent from the subject prior to participation in any study-related procedures if the subject is 18 years of age or older, or from the legally authorized representative/guardian if the subject is under 18 years of age.
8. Must have the signature of the subject on the assent form, as required by Institutional Review Board (IRB) guidelines, if the subject is under 18 years of age.

Exclusion Criteria:

1. Suspected viral or allergic conjunctivitis or suspected fungal or acanthamoeba infections at Screening in either eye.
2. Suspected iritis/uveitis or episcleritis/scleritis at Screening in either eye or history of either condition.
3. Active ulcerative keratitis, specifically any epithelial loss greater than punctate keratitis (eg, confluent epithelial loss or any subepithelial infiltration) in either eye.
4. History of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome in study eye.
5. Uncontrolled systemic or debilitating disease (eg, cardiovascular disease, hypertension, diabetes, or cystic fibrosis) in the opinion of the Investigator.
6. Subjects who are immunocompromised (eg, HIV-positive); any use of immunosuppressive therapy (including chemotherapy).
7. Any use of topical ophthalmic medications, including tear substitutes, within 2 hours before Screening and throughout the study period in either eye.
8. Use of topical ophthalmic antimicrobial therapy within 48 hours prior to Screening. Use of topical ophthalmic antimicrobial therapy other than study medication is prohibited throughout the study period in either eye.
9. Use of topical ophthalmic anti-inflammatory agents (eg, nonsteroidal anti-inflammatory drugs [NSAIDs] or steroids, including steroid-antibiotic combinations) within 48 hours prior to Screening and throughout the study period.
10. Use of systemic antimicrobial therapy for active respiratory tract, urinary tract, skin/soft tissue, or otitis media infection within 72 hours prior to Screening and throughout the study period. Use of a topical dermatologic antibiotic is permitted.
11. Use of systemic steroids within 14 days of screening and throughout the study period. Inhaled, intranasal, and topical dermatological steroids are permitted.
12. Contact lens wear during the study period in study eye. (contact lens wear in an untreated fellow eye is allowed).
13. Ocular surgery (nonlaser or laser) within 6 weeks prior to Screening in study eye.
14. Pregnancy or lactation.
15. Participation in an ophthalmic drug or device research study within 30 days prior to Screening in either eye.
16. Known hypersensitivity to vancomycin, petrolatum, or mineral oil

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Paramount, California
  - Petaluma, California
  - Rancho Cordova, California
  - Deerfield Beach, Florida
  - Waterloo, Iowa
  - Newton, Kansas
  - Pittsburg, Kansas
  - Shawnee Mission, Kansas
  - Havre de Grace, Maryland
  - St Louis, Missouri
  - Asheville, North Carolina
  - High Point, North Carolina
  - Cincinnati, Ohio
  - Roseburg, Oregon
  - Spartanburg, South Carolina
  - Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vancomycin 1.1% | Placebo
Started | 152 | 151
Completed | 149 | 147
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin 1.1% | Placebo | Total
Number analyzed (Participants) | 152 | 151 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (23.69) | 31.9 (26.73) | 31.7 (25.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 83 | 178
  Male | 57 | 68 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 39 | 76
  Not Hispanic or Latino | 115 | 112 | 227
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 8 | 14 | 22
  White | 134 | 124 | 258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 152 | 151 | 303

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinical Resolution of Bacterial Conjunctivitis
Description: Between-group difference in clinical resolution of bacterial conjunctivitis (defined as absence of conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection) at Day 8
Time Frame: 8 days
Population: Modified Intention to Treat population defined as all subjects with Gram positive bacterial conjunctivitis
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin 1.1% | Placebo
Number analyzed (Participants) | 83 | 76
Participants | 71 | 59
Statistical Analysis 1: Comparison: Vancomycin 1.1% vs Placebo; Test type: Superiority; p = 0.2219, Chi-squared

2. Secondary Outcome: Number of Subjects That Display Microbial Eradication
Description: Between-group difference in microbial eradication (absence of all Gram-positive bacterial species present at or above the pathological threshold at baseline) at Day 8
Time Frame: 8 days
Population: modified Intention to Treat population defined as all randomized subjects with Gram positive bacterial conjunctivitis
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin 1.1% | Placebo
Number analyzed (Participants) | 81 | 74
Participants | 56 | 43
Statistical Analysis 1: Comparison: Vancomycin 1.1% vs Placebo; Test type: Superiority; p = 0.1817, Chi-squared

ADVERSE EVENTS:
Time Frame: 8 days of treatment
Arm/Group | Vancomycin 1.1% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/152 | 1/151
Other Adverse Events (participants affected / at risk) | 5/152 | 16/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin 1.1% (N=152) | Placebo (N=151)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin 1.1% (N=152) | Placebo (N=151)
Dry eye (Eye disorders) | 0 (0) | 2 (4)
Punctate keratitis (Eye disorders) | 2 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT02432807/Prot_SAP_000.pdf